CLINICAL TRIAL: NCT03670654
Title: The Effects of an Exercise Program With Pilates Method on Quality of Life and Clinical Control in Asthmatic Patients: a Randomized Controlled Trial
Brief Title: Effects of Pilates Exercises in Asthmatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPEAP
Record Dates: First submitted 2018-09-04; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: Asthma; Exercise; Pilates; Quality of life; Clinical control
MeSH Terms: conditions — Asthma; Motor Activity | interventions — Exercise Movement Techniques; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All the measurements will be performed by a blinded professional, who will be masked from randomization and other results. For each test, the same investigator will be maintained before and after the intervention. The participants will know what treatment (exercise) they will receive, but they don't will know what exercise belongs to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Method (Active Comparator): The intervention of active comparator will be Pilates Method exercises.
  Interventions: Other: Pilates
- Muscle stretching exercises (Sham Comparator): The intervention of sham comparator will be muscle stretching exercises.
  Interventions: Other: Muscle stretching

INTERVENTIONS:
Other: Pilates — The Pilates exercises will be performed in 12 weeks with 40-minute sessions, three times a week: 2 at ambulatory and 1 at home. Ambulatory sessions will be supervised by a physical therapist in non-consecutive days. Patients could be grouped in classes with a maximum of 4 subjects. The first two weeks will be spent learning the technique and, in the third week, patients will receive an exercise booklet for in-home training. Will be used the classical solo Pilates exercises, adapted for non-trained individuals. Before and after each session, patients will be evaluated in relation to expiratory peak flow, blood pressure, heart rate and asthma symptoms.
  Arms: Pilates Method
Other: Muscle stretching — The muscle stretching exercises will be performed in 12 weeks with 40-minute sessions, three times a week: 2 at ambulatory and 1 at home. Ambulatory sessions will be supervised by a physical therapist in non-consecutive days. Patients could be grouped in classes with a maximum of 4 subjects. Patients will practice muscle stretching exercises for principal muscle groups, performed with 3 repetitions, 15 seconds sustain and 1 minute interval. Before and after each session, the patients will be evaluated in relation to expiratory peak flow, blood pressure, heart rate and asthma symptoms.
  Arms: Muscle stretching exercises

SUMMARY:
Asthma is a chronic respiratory disease with high prevalence worldwide, considered an important cause of morbidity, mortality and high economic costs. Aerobic physical exercise has great merit as non-pharmacological treatment and other exercise modalities have being studied. However, there are few data in the literature about the effects of Pilates method in patients with asthma. The objective of this study is evaluate the effects of a program of exercise using Pilates on health factors related to quality of life in patients with moderate or severe persistent asthma. Patients will be also evaluated about disease control, anxiety and depression symptoms, functional capacity, lung function, respiratory muscle strength, thoracoabdominal mechanics and level of daily life physical activity. The investigators' hypothesis is that strengthening of the deep trunk muscles promotes a mechanical fixation of the thorax, contributing to the clinical improvement of patients with asthma.

DETAILED DESCRIPTION:
This is a randomized, controlled and single blinded trial. Thirty adults with moderate or severe persistent asthma will be randomly assigned into two groups: Pilates method - PM (training group) or muscle stretching exercises - MSE (control group). All subjects will receive the same educational session and will perform the physical exercise proposed for the group for 12 weeks, 3 times/week, 40-minute sessions. The data normality will be analyzed by Kolmogorov-Smirnov, the variables obtained before interventions will be compared with the Student t-test or Mann-Whitney U-test. Comparisons of the initial and final data on outcomes will be analyzed with repeated measures ANOVA with appropriate post hoc of Holm-Sidak. The significance level will be set to 5% for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Asthma moderate and severe
* Asthma will diagnosed (Global Initiative for Asthma -GINA)
* Asthma medication according recommendations from GINA
* Body Mass Index ≥18.5 kg/m2 and <35 kg/m2
* Sedentary
* Medical treatment, for at least 6 months
* Clinically stable (i.e., no exacerbation or medication changes for at least 30 days)

Exclusion Criteria:

* Current or ex-smokers (who have given up smoking less than 1 year and/or tobacco charge greater than 10 pack-years)
* Cardiovascular, musculoskeletal and other chronic lung diseases
* Pregnant
* Active cancer
* Uncontrolled hypertension or diabetes
* Continuous use of oral corticosteroid
* Psychiatric disease or cognitive deficit

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-14 (Estimated)

PRIMARY OUTCOMES:
Change in health related quality of life | Change from baseline after 3 months of intervention
  Health related quality of life will be assessed by Asthma Quality Life Questionnaire (AQLQ). The AQLQ is composed by 32 items rated on a 7-point scale ranging from 7 = without limitation to 1 = maximum limitation and grouped in 4 domains: activity limitations (11 items), symptoms (12 items), emotional function (5 items) and environmental stimuli (4 items). Total score will be obtained by the average of the 32 items. The score of each domain will be obtained by the average of the items that compose the domain. A higher score indicates a better quality of life in relation asthma disease and a minimal important difference of 0.5 points results in clinically improvement or deterioration for total score and for each domain.

SECONDARY OUTCOMES:
Change in clinical control | Change from baseline after 3 months of intervention
  Clinical control will be evaluated by asthma control questionnaire (ACQ). The ACQ consists of 7 items rated on a 7-point scale ranging from 0 = without limitation to 6 = maximum limitation and the score will be obtained by the average of the items. A higher score indicates worse control and a change of 0.5 point after intervention is clinically important. Asthma will be considered as controlled (ACQ <0.75 points), not well controlled and poorly controlled asthma (ACQ >1.5 points).
Change in the level of anxiety and depression | Change from baseline after 3 months of intervention
  The symptoms of anxiety and depression will be assessed by Hospital Anxiety and Depression Scale (HADS). The scale is composed by 14 items divided into 2 subscales, each containing 7 items. Each item was scored from 0 to 3, with a maximum score of 21 points for each subscale. The score of each subscale will be obtained by summing the items.
Change in thoracoabdominal mechanics | Change from baseline after 3 months of intervention
  The thoracoabdominal mechanics will be assessed by optoelectronic plethysmography
Change in respiratory muscle strength | Change from baseline after 3 months of intervention
  The strength of the respiratory muscles will be assessed by manovacuometry
Change in pulmonary function | Change from baseline after 3 months of intervention
  Lung volumes will be assessed by Spirometry
Change in functional capacity | Change from baseline after 3 months of intervention
  The functional capacity will be assessed by the Incremental Shuttle Walking Test (ISWT)
Change in daily life physical activity | Change from baseline after 3 months of intervention
  Daily life physical activity will be assessed using an accelerometer (actigraph activity monitor)

OTHER OUTCOMES:
Change in anthropometric dates | Change from baseline after 3 months of intervention
  The body mass index (BMI) will be calculated by the ration between weight in kilograms and height in meter squared (kg/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinical Hospital of São Paulo University medical school (HCFMUSP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No